CLINICAL TRIAL: NCT03994406
Title: A Controlled Phase 2 Study for Prolongation of Contact Lens Comfortable Wear Duration by CLM2 Topical Gel
Brief Title: Prolongation of Contact Lens Comfortable Wear Duration by CLM2 Topical Gel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glia, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLM-1
Record Dates: First submitted 2019-06-20; First posted 2019-06-21 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Contact Lens Discomfort; Contact Lens-induced Corneal Disorder; Contact Lens Acute Red Eye; Contact Lens-induced Corneal Fluorescein Staining
Keywords: contact lens; ocular erythema; contact lens discomfort

STUDY DESIGN:
Intervention Model Description: 1:1, study drug:placebo; block design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: 3-digit randomized number assignment with matching by age within 10 years, and within 5 years of lens wear. Study drug:placebo, 1:1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CLM2 Topical Gel (Experimental): CLM2 topical gel to be applied dermally to forehead twice daily, in the morning and at bedtime.
  Interventions: Drug: CLM2 topical gel
- Placebo Topical Gel (Placebo Comparator): Placebo topical gel to be applied dermally to forehead twice daily, in the morning and at bedtime.
  Interventions: Drug: Placebo topical gel

INTERVENTIONS:
Drug: CLM2 topical gel — Active topical gel for forehead dermal application
  Arms: CLM2 Topical Gel
Drug: Placebo topical gel — Placebo topical gel for forehead dermal application
  Arms: Placebo Topical Gel

SUMMARY:
This study compares contact lens comfortable wear duration, and signs and symptoms of contact lens discomfort, test versus control.

DETAILED DESCRIPTION:
The clinical hypothesis is that CLM2 topical gel applied dermally on the forehead twice daily will be more effective than placebo (a) in reducing or eliminating ocular discomfort associated with contact lens wear, (b) prolong hours of comfortable wear, (c) prolong total hours of contact lens wear, (d) improve ease of insertion and removal of contact lens, and ( c) reduces friction between cornea/lens and lens/eyelid, without use of artificial eye drops or gels. One mechanism supporting this hypothesis is preliminary evidence of increased meibum secretion following CLM2 topical gel application.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of any race ≥18 years of age at Visit 1 Screening.
2. Has provided verbal and written informed consent.
3. Be able and willing to follow instructions, including participation in all study assessments and visits.
4. Has been wearing soft contact lens in both eyes at least 2 days per week for at least a month.
5. Duration of comfortable lens wear daily is less than desired.
6. Suffers from at least two other symptoms while wearing lens with contact lens discomfort of grade 2 or higher:

   1. Dryness.
   2. Grittiness
   3. Blurred vision
   4. Itching
   5. Conjunctival redness
   6. Burning
   7. Stinging.
   8. Lens awareness
   9. Use of artificial tears or gels two or more times a day during contact lens wear hours.
7. Berkeley Dry Eye Flow Chart (DEFC) score ≥3.

Exclusion Criteria:

1. BCVA at baseline <20/40.
2. Wearing contact lens only in one eye.
3. Wearers of the following contact lenses: Extended wear, prosthetic, scleral, and intracorneal gas permeable.
4. Pregnant women or women of childbearing potential who are not using contraception.
5. Diagnosis of the following autoimmune diseases: Addison's disease, Grave's disease, Hashimoto's thyroiditis, lupus, and Sjogren's syndrome.
6. Comorbidity with other severe or chronic eye conditions that in the judgment of the investigator will interfere with study assessments, such dystrophies, infections, etc.
7. Has a condition or be in a situation that, the opinion of the investigator, that may interfere significantly with the subject's participation in the study. No active ocular condition or disease.
8. Has a known adverse reaction and/or sensitivity to either study drug or its components.
9. Unwilling to remove contact lens overnight.
10. Unwilling to attempt to wear contact lens seven (7) days a week during the study period.
11. Plan to change brand of contact lens during study period.
12. Unwilling to wear contact lens for at least 10 hours if comfort permits, or until discomfort requires removal of contact lens prior to 10 hours.
13. Unwilling to discontinue swimming with immersed head for the duration of the study.
14. Unwilling to withhold the use of artificial tears, gels, or wetting agents during periods when contact lens is worn during the study period.
15. Cannot withhold the following medications during the study period:

    antihistamines, some diuretics, antidepressants, antipsychotics, Restasis, Xiidra, Accutane, glaucoma medications, other anti-cholinergics; as well as gabapentin.
16. Currently enrolled in an investigational drug or device study or have used an investigational drug or device within 30 days prior to Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Hours of continuous comfortable contact lens wear | 21 days
  Change in total hours per day
Contact Lens Questionnaire-8 (CLDEQ-8) | 21 days
  Change in total score (0-37 worst)
Berkeley Dry Eye Flow Chart | 21 days
  Change in grade (1-5 worst)
Fluorescein corneal staining | 21 days
  Change in score (0-3 worst)

SECONDARY OUTCOMES:
Eye discomfort from CLDEQ-8, frequency | 21 days
  Change in score (0-4 worst)
Eye discomfort from CLDEQ-8, intensity | 21 days
  Change in score (0-5 worst)
Glia contact lens symptoms questionnaire | 21 days
  Change in total score (0-64)
Fluorescein conjunctival staining | 21 days
  Change in conjunctival staining (0-3 worst)
Tear film examination by TearScan | 60-80 minutes
  Change in total score (0-3 best)
Tear film examination by TearScan | 21 days
  Change in total score (0-3 best)
Tear film breakup time | 60-80 minutes
  Change in score (seconds)
Tear film breakup time | 21 days
  Change in score (seconds)
Tear meniscus height | 60-80 minutes
  Change in height (mm)
Tear meniscus height | 21 days
  Change in height (mm)
Visual acuity | 21 days
  Change in visual acuity
Tear osmolarity | 21 days
  Change in tear osmolarity (mOsm/L)
Schirmer test | 21 days
  Change in wetting length (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Meng C. Lin, OD,PhD,FAAO, Principal Investigator — University of California, Berkeley
Locations (1):
- UC Berkeley Clinical Research Center, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: No